CLINICAL TRIAL: NCT00016172
Title: A Phase I Study of ZD0473 and Doxil in Patients With Advanced Refractory Cancer
Brief Title: ZD0473 and Doxorubicin in Treating Patients With Advanced Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 00-044; CDR0000068603 (Registry Identifier: PDQ (Physician Data Query)); NCI-G01-1942
Record Dates: First submitted 2001-05-06; First posted 2004-02-16 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Lymphoma; Small Intestine Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; small intestine lymphoma; unspecified adult solid tumor, protocol specific; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; primary central nervous system non-Hodgkin lymphoma; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; intraocular lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Intraocular Lymphoma; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — amminedichloro(2-methylpyridine)platinum(II)

INTERVENTIONS:
Drug: pegylated liposomal doxorubicin hydrochloride
Drug: picoplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase I trial to study the effectiveness of combining ZD0473 and doxorubicin in treating patients who have advanced solid tumors or lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of ZD0473 and doxorubicin HCl liposome in patients with advanced or metastatic solid tumors or lymphoma. II. Determine the qualitative and quantitative toxic effects of this regimen in this patient population. III. Determine the pharmacokinetics of these drugs in this patient population. IV. Determine the antitumor activity of this regimen in this patient population.

OUTLINE: This is a dose-escalation study. Patients receive doxorubicin HCl liposome IV over 60 minutes followed by ZD0473 IV over 60 minutes on day 1. Treatment repeats every 28 days for a maximum of 6 courses in the absence of disease progression or unacceptable toxicity. Patients with partial response (PR) or complete response (CR) may continue treatment until disease progression or until 2 courses after maximum response. Cohorts of 3-6 patients receive escalating doses of doxorubicin HCl liposome and ZD0473 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 3 or 3 of 6 patients experience dose-limiting toxicity. Patients are followed at 4 weeks and 3 months. Patients with PR or CR ongoing continue follow-up every 3 months until relapse.

PROJECTED ACCRUAL: Approximately 24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed advanced or metastatic solid tumors or lymphoma Refractory to standard curative therapy OR No curative therapy exists Serologically, clinically, and/or radiographically assessable disease No newly diagnosed brain metastases Intracranial disease that is stable for at least 6 months allowed

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than upper limit of normal (ULN) AST or ALT no greater than 2.0 times ULN Alkaline phosphatase no greater than 2.0 times ULN Renal: Creatinine no greater than ULN Creatinine clearance at least 60 mL/min Cardiovascular: Ejection fraction at least 50% Other: No underlying medical condition that would preclude study or that is uncontrolled No active serious infection No neurotoxicity or preexisting grade 3 or higher neuropathy Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 5 days since prior immunotherapy Chemotherapy: At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas and similar compounds) No more than 3 prior chemotherapy regimens for metastatic disease No prior anthracycline exposure exceeding 300 mg/m2 doxorubicin No prior doxorubicin HCl liposome Endocrine therapy: At least 5 days since prior hormonal therapy Radiotherapy: At least 3 weeks since prior radiotherapy and recovered No prior radiotherapy to more than 30% of functioning bone marrow Surgery: At least 3 weeks since prior major surgery Other: No other concurrent experimental drugs No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-11; Primary Completion 2002-04 (Actual); Study Completion 2002-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R. Spriggs, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States